CLINICAL TRIAL: NCT02879643
Title: A Pilot Study of Vincristine Sulfate Liposome Injection (Marqibo®) in Combination With UK ALL R3 Induction Chemotherapy for Children, Adolescents, and Young Adults With Relapse of Acute Lymphoblastic Leukemia
Brief Title: Vincristine Sulfate Liposome Injection (Marqibo®) in Combination With UK ALL R3 Induction Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2012-002
Record Dates: First submitted 2016-08-16; First posted 2016-08-26 (Estimated); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2022-07

CONDITIONS: ALL, Childhood; Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Leukemia, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Marqibo and UK ALL R3 backbone (Experimental): * Marqibo®: given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Interventions: Drug: Marqibo
- Cohort B: Marqibo and lower intensity UK ALL R3 backbone (Experimental): * Marqibo®: given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Interventions: Drug: Marqibo
- Cohort C: Marqibo and maintenance regimen (Experimental): * Marqibo®: given by intravenous (IV) infusion on day 1
  * Dexamethasone orally twice daily on days 1-5
  * Methotrexate: given orally on days 1 and 8
  * Mercaptopurine: given orally daily on days 1-13
  Interventions: Drug: Marqibo

INTERVENTIONS:
Drug: Marqibo — The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.

SUMMARY:
This is a pilot study utilizing Marqibo® (vincristine sulfate liposome injection) combined with dexamethasone, mitoxantrone and asparaginase (UK ALL R3) for relapsed acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This study will utilize Marqibo® as a replacement for standard vincristine in combination with chemotherapy for children with relapsed ALL. The hypothesis is that the incorporation of Marqibo® with combination chemotherapy will be safe and feasible. In the context of this pilot study, overall outcomes and efficacy will be a secondary objective. It is hypothesized that data from this combination may show improved efficacy including, complete remission (CR), minimal residual disease (MRD) negativity, and progression free survival (PFS) rates and safety (i.e., neurotoxicity) in comparison to outcomes in historical regimens, including the UK ALL R3 with standard vincristine.

ELIGIBILITY:
Inclusion Criteria

Age

-Patients must be ≥ 1 and ≤ 21 years of age at the time of enrollment.

Diagnosis

* Cohort A: Patients must have a diagnosis of acute lymphoblastic leukemia (ALL) or mixed phenotypic acute leukemia with ≥ 5% blasts in the bone marrow (M2 or M3), with or without extramedullary disease) or a diagnosis of lymphoblastic lymphoma.
* Cohorts B & C: Patients must have a diagnosis of acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma, or mixed phenotypic acute leukemia with any level of detectable disease (minimal residual disease level acceptable) with or without extramedullary disease

Performance Level -Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age.

Prior Therapy

* Patients must have recovered from the acute toxic effects (≤ Grade 2 or baseline) of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study, unless otherwise specified. Subjects with disease related cytopenias will be eligible.
* Patients must have relapsed or refractory disease after attaining at least a first remission. They may be in first to third relapse..
* Patients with Philadelphia chromosome t(9;22) positive disease must have received at least two prior tyrosine kinase inhibitors.
* Patients who have experienced their relapse after a Hematopoietic stem cell transplantation (HSCT) are eligible, provided they have no evidence of graft-versus-host disease (GVHD) and are at least 100 days post-transplant at the time of enrollment.
* Prior anthracycline lifetime cumulative exposure: Patients must have less than 320 mg/m2 (or 400 mg/m2 if prior cardioprotection) lifetime exposure of anthracycline chemotherapy.

  1. Cohort A: Patients must have less than 320 mg/m2 (or 400 mg/m2 if prior cardioprotection) lifetime exposure of anthracycline chemotherapy (See Appendix 2 for anthracycline calculation worksheet).
  2. Cohorts B & C: There is no limit on prior anthracycline exposure.
* Hematopoietic growth factors: It must have been at least seven days since the completion of therapy with granulocyte colony-stimulating factor (GCSF) or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).
* Biologic anti-neoplastic agents: At least seven days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond seven days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair or vice chair.
* Monoclonal antibodies: At least three half-lives (or 30 days-whichever is longer) of the antibody must have elapsed after the last dose of monoclonal antibody. (e.g., Rituximab = 66 days, Epratuzumab = 69 days)
* Immunotherapy: At least 30 days after the completion of any type of immunotherapy, e.g. tumor vaccines, chimeric antigen receptor T-cells.
* Recent prior chemotherapy: At least 10 days after standard vincristine and the completion of any type of chemotherapy induction regimen. At least 3 weeks after radiation therapy. At least 30 days after the completion of any investigational neoplastic agent is also required. An investigational agent is defined as any drug that is not approved and licensed for sale by the FDA for institutions in the United States, by Health Canada for institutions in Canada and by The Therapeutic Goods Administration for institutions in Australia.

Exceptions:

* There is no time restriction in regard to prior intrathecal chemotherapy provided there is complete recovery from any acute toxic effects of such; it is allowable to enroll a patient that has received IT Cytarabine (ARA-C), IT Methotrexate (MTX) or triple IT therapy within 14 days of enrollment as part of their evaluation to diagnose disease relapse. The IT therapy given within 14 days of initiation of protocol specified chemotherapy, may substitute for the day 1 IT in cohorts A and B
* Subjects with rapidly progressive disease may receive hydroxyurea until they begin study therapy;
* Patients who relapse while on maintenance-type ALL therapy or are receiving maintenance therapy for disease stabilization will not require a wash-out period before entry into this study. However, there must be at least 10 days after any dose of standard vincristine.

Renal and Hepatic Function

* Renal function: Patient's serum creatinine must be ≤ 1.5 x institutional upper limit of normal (ULN) according to age. If the serum creatinine is greater than 1.5 times normal, the patient must have a calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70milliliter/min/1.73m2. Alternatively, a 24-hour creatinine clearance may also be used.
* Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be < 5 x institutional upper limit of norm ULN. Total bilirubin must be ≤ 1.5 x ULN (except in the case of subjects with documented Gilbert's disease ≤ 5 × ULN).

Cardiac Function

-Patients must have a shortening fraction ≥ 27% or an ejection fraction ≥ 55% by echocardiogram, cardiac MRI or multigated acquisition scan (MUGA).

Reproductive Function

* Female patients must not be pregnant and those of childbearing potential must have a negative urine or serum pregnancy test confirmed within one week prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of childbearing potential must agree to use an effective method of contraception during the study.

Exclusion Criteria

Patients will be excluded if they have isolated testicular disease.

Patients will be excluded if they have previously received Marqibo®.

Patients will be excluded if they have a known allergy to any of the drugs used in the study, with the exception that patients with an allergy to PEG-asparaginase who can receive Erwinia asparaginase are eligible. Patients unable to receive any formulation of asparaginase may only enroll on cohort C

Patients will be excluded if they have active, uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment.

Patients who require azole antifungal agents will be excluded. Azoles must be discontinued at least one week prior to the start of Marqibo®.

Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, another investigational agent or immunotherapy during the study period.

Patients with pre-existing, persistent grade 2 or greater sensory or motor neuropathy from any cause will be excluded.

Patients will be excluded if they have, significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or adherence with the protocol treatment or procedures or interfere with consent, study participation, follow up, or interpretation of study results.Patients with Down syndrome will not be eligible for enrollment on Cohort A

Patients with a known history of human immunodeficiency virus (HIV) will will be excluded due to the increased risk of complications such as severe infection and unknown interaction of Marqibo® with antiretroviral drugs.

Active hepatitis B or C infection as defined by seropositive for hepatitis B (hepatitis B surface antigen (HBsAg)) or hepatitis C and elevated liver transaminases (defined as above the ULN per the institution normal ranges).

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (28):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - UCSF School of Medicine, San Francisco, California
  - The Children's Hospital, University of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - National Cancer Institute, Pediatric Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Cancer Center, Baylor, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Lady Cilento Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Parkville, Victoria
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - Sainte-Justine University Hospital Center, Montréal, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shah NN, Schafer ES, Chi YY, Malvar J, Heym KM, Place AE, Burns M, Chang BH, Slone T, Verma A, Gossai N, Shaw PH, Burke MJ, Hermiston M, Schore RJ, Cooper T, Pauly M, Rushing T, Jarosinski P, Florendo E, Yates B, Widemann BC, Peer CJ, Figg WD, Silverman LB, Bhojwani D, Wayne AS. Vincristine Sulfate Liposome Injection With Combination Chemotherapy for Children, Adolescents, and Young Adults With Relapsed Acute Lymphoblastic Leukemia: A Therapeutic Advances in Childhood Leukemia and Lymphoma Consortium Trial. Pediatr Blood Cancer. 2025 May;72(5):e31584. doi: 10.1002/pbc.31584. Epub 2025 Feb 12. PMID 39937083

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone: * Marqibo® (1.5 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort A Dose Level 2: Marqibo and UKALL R3 Backbone: Marqibo® (2.0 mg/m^2): given byintravenous (IV)infusion on days 1, 8,15 and 22. Dexamethasone orallytwice daily on days 1-5and 15-19. Mitoxantrone: given byintravenous (IV)infusion on days 1 and2. PEG-asparaginase:given as an injectioninto the muscle on says3 and 17. Methotrexate IT: givenintrathecally (used totreat the brain andspinal cord and is givenusing a needle insertedinto the spinal canal) ondays 1 and 8.
  Marqibo: The focus of thestudy design and statisticalanalysis is to determinewhether Marqibo® can besubstituted for standardvincristine and successfullyadministered to patients withrelapsed ALL in threedifferent treatment cohorts:(A) treatment with the UK ALLR3 regimen; (B) treatmentwith UK ALL R3 regimenwithout mitoxantrone, and (C)treatment with ALLmaintenance therapy.Secondary objectives includeestimating rates of serioustoxicities and therapy delaysin each of these cohorts.
- Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone: * Marqibo® (1.5 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort B Dose Level 2: Marqibo and LowerIntensity UK ALL R3Backbone: Marqibo® (2.0 mg/m^2): given byintravenous (IV)infusion on days 1, 8,15 and 22. Dexamethasone orallytwice daily on days 1-5and 15-19. PEG-asparaginase:given as an injectioninto the muscle on days3 and 17. Methotrexate IT: givenintrathecally (used totreat the brain andspinal cord and is givenusing a needle insertedinto the spinal canal) ondays 1 and 8.
  Marqibo: The focus of thestudy design and statisticalanalysis is to determinewhether Marqibo® can besubstituted for standardvincristine and successfullyadministered to patients withrelapsed ALL in threedifferent treatment cohorts:(A) treatment with the UK ALLR3 regimen; (B) treatmentwith UK ALL R3 regimenwithout mitoxantrone, and (C)treatment with ALLmaintenance therapy.Secondary objectives includeestimating rates of serioustoxicities and therapy delaysin each of these cohorts.
- Cohort C Dose Level 2: Marqibo and Maintenance Regimen: * Marqibo®(2.0 mg/m^2): given by intravenous (IV) infusion on day 1
  * Dexamethasone orally twice daily on days 1-5
  * Methotrexate: given orally on days 1 and 8
  * Mercaptopurine: given orally daily on days 1-13
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
Period: Overall Study
Arm/Group | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone | Cohort A Dose Level 2: Marqibo and UKALL R3 Backbone | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort B Dose Level 2: Marqibo and LowerIntensity UK ALL R3Backbone | Cohort C Dose Level 2: Marqibo and Maintenance Regimen
Started | 12 | 4 | 6 | 2 | 5
Completed | 12 | 4 | 5 | 1 | 5
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone: * Marqibo® (2.0 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone: * Marqibo® (2.0 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort C Dose Level 2: Marqibo and Maintenance Regimen: * Marqibo® (2.0 mg/m^2): given by intravenous (IV) infusion on day 1
  * Dexamethasone orally twice daily on days 1-5
  * Methotrexate: given orally on days 1 and 8
  * Mercaptopurine: given orally daily on days 1-13
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Total: Total of all reporting groups
Arm/Group | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone | Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort C Dose Level 2: Marqibo and Maintenance Regimen | Total
Number analyzed (Participants) | 12 | 4 | 6 | 2 | 5 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 4 | 5 | 2 | 4 | 27
  Between 18 and 65 years | 0 | 0 | 1 | 0 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 12.3 [1.8 to 17.3] | 8.7 [5 to 14.4] | 12 [8.2 to 19.6] | 12.7 [8.9 to 16.8] | 15.8 [4 to 19.5] | 12.4 [1.8 to 19.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 1 | 2 | 12
  Male | 7 | 3 | 3 | 1 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 10 | 2 | 4 | 2 | 2 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 | 4 | 6 | 2 | 5 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities as a Measure of Safety and Tolerability
Description: Number of Participants with Dose Limiting Toxicities as a Measure of Safety and Tolerability at different dose levels of Marqibo. Dose Level 1 = 1.5 mg/m^2. Dose Level 2 = 2.0 mg/m^2. Cohort A and B accrued at both Dose Levels. Cohort C accrued only at Dose Level 2.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone: * Marqibo®(1.5 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone: * Marqibo®(2.0 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone: * Marqibo®(1.5 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone: * Marqibo®(2.0 mg/m^2): given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
Arm/Group | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone | Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort C Dose Level 2: Marqibo and Maintenance Regimen
Number analyzed (Participants) | 12 | 4 | 6 | 2 | 5
Participants
  DLT | 0 | 2 | 0 | 1 | 0
  No DLT | 12 | 2 | 6 | 1 | 5

ADVERSE EVENTS:
Time Frame: Through 30 days after the last day of protocol therapy (cycle 1 only), approximately 9 weeks
Groups:
- Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone; Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone: * Marqibo®: given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * Mitoxantrone: given by intravenous (IV) infusion on days 1 and 2.
  * PEG-asparaginase: given as an injection into the muscle on says 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone; Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone: * Marqibo®: given by intravenous (IV) infusion on days 1, 8, 15 and 22.
  * Dexamethasone orally twice daily on days 1-5 and 15-19.
  * PEG-asparaginase: given as an injection into the muscle on days 3 and 17.
  * Methotrexate IT: given intrathecally (used to treat the brain and spinal cord and is given using a needle inserted into the spinal canal) on days 1 and 8.
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
- Cohort C: Marqibo and Maintenance Regimen: * Marqibo®: given by intravenous (IV) infusion on day 1
  * Dexamethasone orally twice daily on days 1-5
  * Methotrexate: given orally on days 1 and 8
  * Mercaptopurine: given orally daily on days 1-13
  Marqibo: The focus of the study design and statistical analysis is to determine whether Marqibo® can be substituted for standard vincristine and successfully administered to patients with relapsed ALL in three different treatment cohorts: (A) treatment with the UK ALL R3 regimen; (B) treatment with UK ALL R3 regimen without mitoxantrone, and (C) treatment with ALL maintenance therapy. Secondary objectives include estimating rates of serious toxicities and therapy delays in each of these cohorts.
Arm/Group | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone | Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone | Cohort C: Marqibo and Maintenance Regimen
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/6 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 7/12 | 4/4 | 0/6 | 1/2 | 5/5
Other Adverse Events (participants affected / at risk) | 12/12 | 4/4 | 6/6 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone (N=12) | Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone (N=4) | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone (N=6) | Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone (N=2) | Cohort C: Marqibo and Maintenance Regimen (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Encephalitis infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A Dose Level 1: Marqibo and UK ALL R3 Backbone (N=12) | Cohort A Dose Level 2: Marqibo and UK ALL R3 Backbone (N=4) | Cohort B Dose Level 1: Marqibo and Lower Intensity UK ALL R3 Backbone (N=6) | Cohort B Dose Level 2: Marqibo and Lower Intensity UK ALL R3 Backbone (N=2) | Cohort C: Marqibo and Maintenance Regimen (N=5)
Anemia (Blood and lymphatic system disorders) | 11 | 4 | 6 | 2 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 2 | 0 | 1
Blurred vision (Eye disorders) | 1 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 3 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 1 | 2 | 1 | 2
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 3 | 1 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 2 | 1 | 1
Fever (General disorders) | 4 | 1 | 2 | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (General disorders) | 2 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Encephalitis infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 | 3 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 3 | 1 | 1
Alanine aminotransferase increased (Investigations) | 9 | 3 | 4 | 2 | 4
Alkaline phosphatase increased (Investigations) | 4 | 1 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 3 | 5 | 2 | 4
Blood bilirubin increased (Investigations) | 2 | 1 | 3 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 1 | 0 | 0
GGT increased (Investigations) | 3 | 2 | 0 | 0 | 2
INR increased (Investigations) | 1 | 0 | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 8 | 3 | 6 | 2 | 4
Neutrophil count decreased (Investigations) | 9 | 4 | 6 | 2 | 3
Platelet count decreased (Investigations) | 10 | 4 | 5 | 2 | 4
Serum amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight loss (Investigations) | 2 | 0 | 2 | 1 | 0
White blood cell decreased (Investigations) | 9 | 4 | 6 | 2 | 5
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 1 | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 3 | 4 | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 2 | 2 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 4 | 5 | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 1 | 5 | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 4 | 3 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 2 | 4 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 10 | 4 | 4 | 1 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 2 | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 2 | 1 | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 4 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT02879643/Prot_SAP_ICF_000.pdf